CLINICAL TRIAL: NCT03218956
Title: Determination of Dietary Protein Requirements in Healthy Women During Stages of Lactation
Brief Title: Protein Requirement During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Principal investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H17-00079
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy
Keywords: Protein requirement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protein intake (Experimental): Dietary supplement: Protein intake
  Interventions: Dietary Supplement: Dietary supplement: Protein intake

INTERVENTIONS:
Dietary Supplement: Dietary supplement: Protein intake — Oral consumption of houly experimental meals. Includes 4 meals containing a mixture of free amino acids, carbohydrates from a flavored liquid, fat from corn oil and protein free cookies.
  The last 4 meals will in addition contain labelled labelled 13C phenylalanine.

SUMMARY:
It is well established that a breast-feeding women need more protein in their diet compared to non-lactating women, but how much additional protein is needed remains unclear. There is reason to believe that the current Dietary Reference Intake (DRI) recommendations for breast-feeding women are too low. To gain better understanding, we plan to study healthy breast-feeding women 20 - 45 yrs, between 3 - 5 months lactation and 6 - 8 months lactation. We will use the indicator amino acid oxidation technique (IAAO), which is a modern, quick and safe research method.

DETAILED DESCRIPTION:
Purpose:

To determine the dietary protein intake requirement in healthy lactating women during the exclusive breast-fed period (3 - 5 months lactation) and during weaning (6 - 8 months lactation).

Hypothesis:

Recent stable isotope-based research using the IAAO technique indicate that current protein intake recommendations are underestimated in adults by ~40 %, in school aged children ~75 % and pregnant women during early and late gestation by ~39 % and ~73 %, respectively.

Therefore we hypothesize that that protein requirements will be increased during both phases of lactation above that of the current recommendations

Justification:

The WHO advocates that all newborn infants are exclusively breast-fed for the first 6 months of life, followed by a period of weaning, with appropriate complementary feeds, which is recommended to continue until the child's second birthday. The period of lactation from the mother's perspective of up to 2 years for each child, represents a considerable period of adult life. Adequate protein intake during lactation is important - if a woman's dietary intake of protein is inadequate, her own lean mass will be depleted to support the growth of the infant. Currently, dietary protein intake recommendations are based on nitrogen balance studies conducted in men and recommendations for breast-feeding women are extrapolated from these studies, and there is little breast-feeding specific data.

Objectives:

To determine the protein requirements during lactation and examine whether protein needs are significantly altered during exclusive breastfeeding (~3 - 5 mo post parturition) and partial breast feeding (~6 - 8 mo post parturition).

Research design:

A minimum of 10 women will be recruited. Each mother will participate in up to 8 study days, 4 during the exclusively breast-fed period and 4 during the partial breast-fed period, for a total of 40 data points (study days) during each lactation period. We hope to retain the same women for all 8 study days to minimize data variability.

Potential participants will meet us for a preliminary assessment where we will evaluate their eligibility to participate in the study. The preliminary assessment will take approximately 1 hour during which we will examine body composition (Bioelectrical impedance, skin-fold measurements, height and weight), resting energy expenditure (by indirect calorimetry) and medical history (questionnaire). We will collect a 3 day food diary, to determine usual food intake and food preferences. Based on the 3 day food record we will prescribe a standardized diet two days prior to the study day to ensure protein intake of 1.5 g/kg/day and 1.7 x resting energy.

During each study day, the participants will randomly receive 1 of 40 test protein intakes. Each subject will participate in one study day at approximately 14, 16, 18, 20 weeks postpartum and 24, 28, 30 and 32 weeks postpartum, respectively, for a total of up to 8 study days.

The test protein intakes will be administered in an experimental diet. The study day diets will consist of 8 isocaloric and isonitrogenic meals provided hourly, each meal presenting 1/12 of the daily energy requirement. Study day diet is composed of a crystalline amino acid mixture based on the composition of egg-protein, flavored with orange Tang, orange Kool-aid crystals and corn oil.

A stable isotope tracer will be added to the 5th - 8th meal. We will measure the rate of oxidation of this tracer expired in breath (F13CO2), and flux of this tracer by its enrichment in urine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy lactating women
* With a healthy baby
* Exclusively breast feeding (3 - 5 months) and are partially breast-feeding women (6 - 8 months) - not supplementing with infant formula

Exclusion Criteria:

* Women below 20 yrs or above 45 yrs of age
* Women who are breast-feeding more than one child
* Women who are not exclusively breast feeding (3 - 5 months) and women who are supplementing with infant formula or have not transitioned to solid foods by 6 - 8 months.
* Women not in good health and have a metabolic, neurological, genetic, or immune disorder.
* Women who are claustrophobic (we will place a clear hood, which can easily be removed, over the participants head for approximately 20 min to measure energy expenditure).
* Women who are substance dependent (i.e. alcohol, cigarette, illicit drugs)
* Women who are allergic to eggs and egg protein
* Women who do not have a healthy baby

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
13C Phenylalanine Oxidation | 8 hours
  Urine, breath and a single blood sample will be collected during the study to measure the rate of oxidation of 13C phenylalanine.

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with other researchers

REFERENCES:
- See also: Abstract — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7257931/